CLINICAL TRIAL: NCT04230785
Title: Clinical Significance of Circulating Non-coding RNA in Acute Ischemic Stroke with Endovascular Treatment (EVTRNA)
Brief Title: Circulating Non-coding RNA in Acute Ischemic Stroke with Endovascular Treatment (EVTRNA)
Acronym: EVTRNA
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: Zhongda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EVTRNA
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Stroke, Acute; Stroke, Ischemic; Endovascular Treatment
Keywords: acute ischemic stroke; noncoding RNA; endovascular treatment; clinical significance; outcome
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples With DNA — An 10 ml peripheral venous blood will be collected from the participants before and after endovascular treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- AIS before EVT group: This group includes patients with acute ischemic stroke (AIS) before endovascular treatment (EVT)
  Interventions: Genetic: Sequencing of circRNA/lncRNA/miRNA
- AIS after EVT group: This group includes patients with acute ischemic stroke (AIS) after endovascular treatment (EVT)
  Interventions: Genetic: Sequencing of circRNA/lncRNA/miRNA

INTERVENTIONS:
Genetic: Sequencing of circRNA/lncRNA/miRNA — Next generation sequencing and quantitative real-time polymerase chain reaction of circular RNA (circRNA), long non-coding RNA (lncRNA) and micro-RNA (miRNA)
  Other Names: Quantitative Real-time polymerase chain reaction

SUMMARY:
EVTRNA is to analyze the differentiated expression pattern of circular RNA (circRNA), long non-coding RNA (lncRNA) and micro-RNA (miRNA) by next-generation sequencing in acute ischemic stroke patients before and/or after endovascular treatment. The candidate circRNA/lncRNA/miRNA will be verified as the biomarker and regulator for progression and prognosis of acute ischemic stroke with endovascular treatment. Further, the candidate non-coding RNA will be used to evaluate the effect of endovascular treatment on both peripheral and central immune after stroke.

DETAILED DESCRIPTION:
Noncoding RNAs have been highlighted to be involved in the pathological process of ischemic stroke (IS). The purpose of this protocol will investigate the differentiated expression pattern of circular RNA (circRNA), long non-coding RNA (lncRNA) and micro-RNA (miRNA) by next-generation sequencing in acute ischemic stroke patients before and/or after endovascular treatment. The candidate circRNA/lncRNA/miRNA will be verified as the biomarker and regulator for progression and prognosis of acute ischemic stroke with endovascular treatment. Further, the candidate non-coding RNA will be used to evaluate the effect of endovascular treatment on both peripheral and central immune after stroke. Distinctive expression patterns of circRNA/miRNA/lncRNA will be identified by the next-generation sequencing and individual quantitative real time polymerase chain reaction (qRT-PCR). A predictive model will be established using logistic regression. The panel of these altered ncRNAs may be associated with the immune status after acute IS and could serve as a regulator for progression and prognosis of acute ischemic stroke with endovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Confirmed acute ischemic stroke by a diffusion-weighted imaging-position lesion on magnetic resonance imaging (MRI) and a new lesion on a brain computed tomography (CT) scan
* Within 24 hours of symptom onset and treat with endovascular therapy
* Good performance status
* Signed an approved informed consents

Exclusion Criteria:

* a history of hemorrhagic infarction, chronic kidney/liver diseases, peripheral arterial occlusive disease, active malignant disease, and inflammatory or infectious diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There will be 5 AIS patients, whose data before and after endovascular treatment will be applied for sequencing the differentiated expression pattern and constraction of diagnosis and predictive models of circRNA/lncRNA/miRNA from the circulating blood. There will be 300 AIS patients, whose data will be applied for validation of such diagnosis and predictive models and investigated the effect of non-coding RNA on immune status after endovascular treatment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Differential expression pattern of circRNA/lncRNA/miRNA in acute ischemic stroke patients before and after endovascular treatment | 90 days
  Differential expression pattern of circular RNA (circRNA), long non-coding RNA (lncRNA) and micro-RNA (miRNA) will be compared in acute ischemic stroke patients before and after endovascular treatment, thus candidate circRNA/lncRNA/miRNA will be verified as biomarkers and regulators for progression and prognosis of acute ischemic stroke with endovascular treatment.

SECONDARY OUTCOMES:
Prognostic value of circRNA/miRNA/lncRNA in acute ischemic stroke with endovascular treatment | 90 days
  The prognosis of AIS patients will be analyzed between differential expressed candidate circRNA/lncRNA/miRNA after they have endovascular treatment.
Correlation of circRNA/lncRNA/miRNA and inflammatory factors in acute ischemic stroke with endovascular treatment | 90 days
  Correlation of circRNA/lncRNA/miRNA and inflammatory factors in acute ischemic stroke before and after endovascular treatment will be explored.
Correlation of circRNA/lncRNA/miRNA and stroke-associated infection | 90 days
  Correlation of circRNA/lncRNA/miRNA and stroke-associated infection will be explored in acute ischemic stroke with endovascular treatment.
Dynamic changes of circRNA/lncRNA/miRNA during the follow-up period | 90 days
  Dynamic changes of circRNA/lncRNA/miRNA will be explored after endovascular therapy during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Junshan Zhou, M.D, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
All information will be available to all researchers
Supporting Information: Study Protocol
Time Frame: All information will be available to all researchers when related investigation has been accepted publicly, and will be available for 5 years.
Access Criteria: All information will be available to all researchers when related investigation has been accepted publicly.

REFERENCES:
- [Background] Deng QW, Li S, Wang H, Sun HL, Zuo L, Gu ZT, Lu G, Sun CZ, Zhang HQ, Yan FL. Differential long noncoding RNA expressions in peripheral blood mononuclear cells for detection of acute ischemic stroke. Clin Sci (Lond). 2018 Jul 31;132(14):1597-1614. doi: 10.1042/CS20180411. Print 2018 Jul 31. PMID 29997237
- Available data/document: Clinical Study Report — http://www.ncbi.nlm.nih.gov/pubmed/?term=Differential+long+noncoding+RNA+expressions+in+peripheral+blood+mononuclear+cells+for+detection+of+acute+ischemic+stroke